CLINICAL TRIAL: NCT04636892
Title: Clinical Correlation of a Novel Wearable Sensor to Detect Cardiovascular Mechanical and Electrical Properties Through Infrasonic Hemodynography
Brief Title: Evaluating Infrasonic Hemodynography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Sanjeev Bhavnani MD, Principal Investigator, Scripps Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-7677
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Aortic Stenosis; Mitral Regurgitation; Pulmonary Hypertension; Heart Failure, Systolic; Cardiovascular Diseases; Coronary Artery Disease
Keywords: infrasonic hemodynography; biomedical device
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Insufficiency; Hypertension, Pulmonary; Heart Failure, Systolic; Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Severe aortic stenosis (Experimental): Patients with echocardiographic evidence of severe aortic stenosis as defined by:
  Aortic Vmax ≥4 m/s or mean ΔP ≥40 mmHg AVA ≤1.0 cm2
  Interventions: Other: MindMics earbud
- Severe mitral regurgitation (Experimental): Patients with echocardiographic evidence of severe mitral regurgitation as defined by:
  * Central jet MR >40% LA or holosystolic eccentric jet MR
  * Vena contracta ≥0.7 cm
  * Regurgitant volume ≥60 mL
  * Regurgitant fraction ≥50%
  * ERO ≥0.40 cm2
  * Angiographic grade 3 to 4+
  Interventions: Other: MindMics earbud
- Heart Failure with Reduced EF <35% (Experimental): Patients with echocardiographic evidence of left ventricular ejection fraction of < or = to 35%
  Interventions: Other: MindMics earbud
- Pulmonary Hypertension (Experimental): Patients with echocardiographic evidence of a mean pulmonary artery pressure (mPAP; supine and at rest) >20mmHg
  Interventions: Other: MindMics earbud
- Suspected coronary artery disease (Experimental): Patients with plan to undergo elective left heart diagnostic catheterization for the assessment of coronary artery disease
  Interventions: Other: MindMics earbud

INTERVENTIONS:
Other: MindMics earbud — Novel noninvasive wearable infrasound sensor

SUMMARY:
This comparative diagnostic accuracy study will determine the accuracy of a noninvasive wearable infrasonic sensor to detect the mechanical, electrical, and hemodynamic function of the cardiovascular system.

DETAILED DESCRIPTION:
This comparative diagnostic accuracy study will determine the accuracy of a noninvasive wearable infrasonic sensor to detect the mechanical, electrical, and hemodynamic function of the cardiovascular system. 25 patients with cardiovascular disease will undergo a comprehensive echocardiogram, electrocardiogram, and cardiac catheterization while wearing a infrasonic earbud device. The infrasonic and hemodynamic waveforms will be analyzed using machine learning with the goal of correlating infrasound data captured by the earbud to the patient's cardiovascular hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Normal Sinus Rhythm
* LV systolic function >53%

Exclusion Criteria:

* 1. Known history of carotid artery disease
* 2. Moderate or greater valvular disease in Group 1
* 3. Other implantable devices (pacemaker, ICD, CardioMems, TENS unit, continuous glucose monitors, etc)
* 4. Active arrhythmia
* 5. Reduced Ejection Fraction (< 35%) other than Group 4
* 6. Hearing loss

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Infrasound Hemodynography | 1 year
  Correlation of Infrasound data to hemodynamic parameter(s) and to cardiac time intervals

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Bhavnani, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Wearable PPG prediction of cardiac output from arterial line measurement in a swine model — https://www.nature.com/articles/s41598-020-74686-6
- See also: Hearables: Multimodal physiological in-ear sensing — https://pubmed.ncbi.nlm.nih.gov/28761162/